CLINICAL TRIAL: NCT01814163
Title: Observational Studies to Explore the Relation Between Angiogenic Markers and the Treatment Response With Carboplatin, Paclitaxel and Bevacizumab in First Line of Advanced Non-small-cell Lung Cancer With Non- Squamous Histology
Brief Title: Observational Post-authorization Studies Carboplatin, Paclitaxel and Bevacizumab
Acronym: ANGIOMET
Status: Completed | Type: Observational
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Other Study IDs: GECP 09-02
Record Dates: First submitted 2012-07-18; First posted 2013-03-19 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Nonsquamous Nonsmall Cell Neoplasm of Lung
Keywords: First line treatment; Non small cell lung cancer, non squamous
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Carboplatin; Bevacizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Paclitaxel, carboplatin and bevacizumab: Paclitaxel 200 mg/m2, carboplatin area under curve (AUC) 6 mg/ml/min plus bevacizumab 15 mg/kg on day 1, every 21 days. Total number of cycles: 6. After 6 cycles bevacizumab on monotherapy until progression
  Interventions: Drug: paclitaxel, carboplatin and bevacizumab

INTERVENTIONS:
Drug: paclitaxel, carboplatin and bevacizumab — Paclitaxel 200 mg/m2, carboplatin area under curve (AUC) 6 mg/ml/min plus bevacizumab 15 mg/kg on day 1, every 21 days. Total number of cycles: 6. After 6 cycles bevacizumab on monotherapy until progression
  Other Names: Taxol, carboplatin, avastin

SUMMARY:
This is a pharmacogenomic study with carboplatin, paclitaxel and bevacizumab as first line therapy in patients with non-squamous advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
This is a observational study prospectively followed post-authorization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should sign inform consent before inclusion in the study that specifies that the clinical treatment entails consent for the analysis of biological samples of tumor and blood.
2. Histologically confirmed diagnosis of advanced non small-cell lung carcinoma, non-squamous cell
3. Patients age 18 years or more
4. Patients will be candidates to received a first line of chemotherapy of carboplatin, paclitaxel and bevacizumab as the best therapeutic option.
5. Evidence of measurable disease per Response Evalutation Criteria in Solid tumors (RECIST)
6. Patients must be avalaible for clinical follow-up
7. Patients with the following hematologic/biochemical values:

   * Absolute Neutrophil Count ANC > 1500/µl.
   * Platelets > 100.000 /µl.
   * Hemoglobine > 10 g/dl.
   * Bilirrubin < 1.5 mg/dl.
   * Aspartate aminotransfereasa (AST) and Alanine transaminase (ALT) ≤ 3 x LSN, except in case of hepatic metastases: upper 5 x LSN
   * Creatinine clearance ≥ 45 ml/min.

Exclusion Criteria:

1. Previous treatment for advanced disease. Chemotherapy is allowed if the initial diagnosis of the patient is limited disease and the patient has received adjuvant or neadjuvant treatment
2. history of haemoptysis (defined as at least half a teaspoon's emission of red blood) in the 3 months prior to inclusion
3. evidence by CT of tumor cavitations, or tumours invading or abutting major blood vessels
4. Known or suspected brain metastases non-treated.
5. Major surgery within 28 days of starting treatment.
6. Minor surgery within 24 hours before starting the treatment.
7. Non-controlled hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg).
8. Patients with coronary disease or uncontrolled arrhytmia, uncontrolled cerebrovascular disease and other clinical conditions that, in judgment of the investigator, contraindicate the patient's participation in the study.
9. History or evidence of bleeding diathesis or hereditary coagulopathy.
10. Contraindication or suspected allergy to the products under investigation in the study:: paclitaxel, carboplatine or bevacizumab.
11. Patients who are pregnant or breasfeeding. Women of childbearing potencial must have a negative pregnancy test performed within 7 days before the onset of treatment.
12. Substance abuse of clinical, psychological or social conditions that can undermine the validity of the informed consent or protocol compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer advanced unresectable, metastatic or recurrent, non-squamous and untreated with chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Correlation between angiogenesis markers and progression free survival. | 1 year

SECONDARY OUTCOMES:
Overal survival | 3 year
Survival at 12 and 24 months | 12-24 months
Objective response | 24 months
Duration of response | 24 months
Treatment security | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bartomeu Massutí, MD, Study Chair — H. Gen. Univ.Alicante; Carlos Camps, MD, Study Chair — H. Gen. Univ. Valencia; Javier de Castro, MD, Study Chair — H. La Paz
Locations (20):
- Spain (20):
  - H. Gen. Universitario Alicante, Alicante, Alicante
  - H. Clínico San Carlos, Madrid, Madrid
  - H. La Paz, Madrid, Madrid
  - H. Gen. Univ. Valencia, Valencia, Valencia
  - Hospital Provincial de Castellón, Castellon
  - Hospital General de Elche, Elche (Alicante)
  - Hospital General de L'Hospitalet, l'Hospitalet (Barcelona)
  - Hospital Insular Gran Canaria, Las Palmas
  - Clínica Quirón, Madrid
  - Fundacion Jiménez Díaz, Madrid
  - Hospital Gregorio Marañon, Madrid
  - Hospital Puerta de Hierro, Majadahonda (Madrid)
  - Clinica Rotger, Palma de Mallorca
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Ntra Sra Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Canarias, Santa Cruz de Tenerife
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Dr. Peset, Valencia
  - Hospital La Fe, Valencia
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- See also: Spanish Lung Cancer Group website — http://www.gecp.org/